CLINICAL TRIAL: NCT06767787
Title: Morbid Obesity and Severe Knee Osteoarthritis - Which Should Be Treated First? A Randomized Cross-over Study
Brief Title: Morbid Obesity and Severe Knee Osteoarthritis - Which Should Be Treated First?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Nick Smith, Dr. Nicholas Smith, Clinical Assistant Professor of Surgery (Orthopaedics), Memorial University of Newfoundland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HREB Application No. 38151
Record Dates: First submitted 2025-01-05; First posted 2025-01-10 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis of Knee; Arthroplasties, Knee Replacement; Sleeve Gastrectomy
Keywords: knee osteoarthritis; bariatric surgery; laparoscopic sleeve gastrectomy; knee replacement; knee arthroplasty; obesity
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity | interventions — Bariatric Surgery; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleeve Gastrectomy then Knee Arthroplasty (Active Comparator): Participants in this arm will undergo laparoscopic sleeve gastrectomy followed by a total knee arthroplasty at least 1 year following the first procedure.
  Interventions: Procedure: laparoscopic sleeve gastrectomy; Procedure: total knee arthroplasty
- Knee Arthroplasty then Sleeve Gastrectomy (Active Comparator): Participants in this arm will undergo total knee arthroplasty followed by laparoscopic sleeve gastrectomy at least 1 year following the first procedure.
  Interventions: Procedure: laparoscopic sleeve gastrectomy; Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — Participants undergoing laparoscopic sleeve gastrectomy (LSG) will be clinically assessed and provided consent to this procedure by one of the bariatric surgeons affiliated with the bariatric surgery program. LSG will be performed at a local tertiary care hospital as either a day procedure or as an overnight stay if medically indicated. Patients will be discharged once they can tolerate a liquid diet. Patients will then attend regular follow-ups with their surgeons and the bariatric surgery program, in accordance with a standardized clinical pathway protocol.
  Other Names: bariatric surgery; sleeve gastrectomy
Procedure: total knee arthroplasty — Patients undergoing unilateral total knee arthroplasty (TKA) will be clinically assessed and provided consent to their procedure by an orthopaedic surgeon trained in joint arthroplasty. TKA will be performed at a local tertiary care hospital as either a day procedure or as an overnight stay if medically indicated. Patients will be discharged once physiotherapy clears them. Patients will attend regular follow-ups with their surgeon in accordance with a standardized clinical pathway protocol.
  Other Names: knee arthroplasty; knee replacement

SUMMARY:
The goal of this study is to determine whether undergoing bariatric surgery before knee replacement leads to better outcomes compared to undergoing knee replacement before bariatric surgery. Our secondary goal is to compare complication rates between these groups to determine if there is a difference based on the order of the two procedures.

Participants will be randomly placed in one of two groups, with each undergoing both procedures but in opposite order. Quality of life will be assessed via questionnaires before and between each procedure, and rates of complications will also be documented to compare their rates between groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI > or = 35, on surgical waitlist for a total knee arthroplasty and laparoscopic sleeve gastrectomy

Exclusion Criteria:

* a history of revision surgery, surgery for neoplastic disease, significant mental illness, ASA class > 3 denoting absence of significant impact of comorbidities, and previous esophagogastric surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
SF-36 Physical Function Component Score | At baseline/enrollment followed by a year following each procedure.
  The 36-Item Short-Form Survey (SF-36) Physical Function Component Score will be assessed 1 year after each procedure as a measure of quality of life.

SECONDARY OUTCOMES:
SF-36 Mental Component Score | At baseline/enrolment followed by a year after each procedure
  The 36-Item Short Form Survey's (SF-36) Mental Component Score will be used to assess participants' quality of life at baseline in addition to after each procedure.
Knee Osteoarthritis Outcome Score (KOOS) | At baseline/enrolment in addition to a year following each procedure
  The KOOS will be used to assess knee-specific function and symptoms at baseline as well as after each procedure.
Post-Operative Outcomes | At 12 and 24 months following each intervention
  Post-operative outcomes following each intervention will be collected, including: hospital bed-day utilization, change in BMI and weight at 12 and 24 months.
Post-Operative Complications | Surveilled every 3 months post- each procedure, until the 12-month postoperative mark.
  Post-operative complications will be surveilled every 3 months following each procedure, including: death from any cause, perioperative or postoperative complications that result in a delay in discharge (e.g., fracture, neurapraxia, sepsis, nosocomial infection, myocardial infarction, bowel obstruction, postoperative nausea & vomiting, venous thromboembolism, cerebrovascular event, and renal failure), wound complications (e.g., infections, hematomas, and dehiscence), prosthetic infection, and unplanned procedures and/or readmission.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - St. Clare's Mercy Hospital, St. John's, Newfoundland and Labrador

IPD SHARING:
Plan to Share IPD: No